CLINICAL TRIAL: NCT04582045
Title: Effect of Prophylactic Negative Pressure Versus Silver Impregnated Silicone Bandage on Cesarean Section Surgical Site Infection Rate
Brief Title: Effect of Prophylactic Negative Pressure Versus Silver Impregnated Silicone Bandage on C-Section Infection Rates
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A180389
Record Dates: First submitted 2020-10-04; First posted 2020-10-09 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2021-12

CONDITIONS: D001458; D011247
Keywords: infection; bandage; cesarean section
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- low risk, silver impregnated: low risk, silver impregnated
  Interventions: Device: silver impregnated dressing
- low risk, border bandage: low risk, border bandage
- high-risk, silver impregnated: high-risk, silver impregnated
  Interventions: Device: silver impregnated dressing
- high-risk, wound vacuum: high-risk, wound vacuum

INTERVENTIONS:
Device: silver impregnated dressing — comparison of Mepilex versus our standard techniques
  Other Names: Mepilex; Wound vacuum
  Groups: high-risk, silver impregnated; low risk, silver impregnated

SUMMARY:
Effect of Prophylactic Negative Pressure versus Silver Impregnated Silicone Bandage on Cesarean Section Surgical Site Infection Rate

DETAILED DESCRIPTION:
Comparison of effect of Prophylactic Negative Pressure versus Silver Impregnated Silicone Bandage on Cesarean Section Surgical Site Infection Rate as compared to wound vacuum in high risk women and traditional border dressing in low risk women in adult women having uncomplicated cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* adult women, pregnant

Exclusion Criteria:

* <18 years old
* surgery complicated by non-routine surgeries (Such as appendectomy)

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: adult women requiring cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 1064 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Goldenberg, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Risk, Border Bandage: low risk, border (traditional) bandage
- High-risk, Wound Vacuum: high-risk, negative-pressure wound vacuum
Period: Overall Study
Arm/Group | Low Risk, Silver Impregnated | Low Risk, Border Bandage | High-risk, Silver Impregnated | High-risk, Wound Vacuum
Started | 446 | 440 | 95 | 83
Completed | 446 | 440 | 95 | 83
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Risk, Border (Traditional) Bandage: low risk, border (traditional) bandage
  standard border wound bandage
- High-risk, Negative-pressure Wound Vacuum: high-risk, negative-pressure wound vacuum
  Commercially available negative-pressure wound vacuum
- Total: Total of all reporting groups
Arm/Group | Low Risk, Silver Impregnated | Low Risk, Border (Traditional) Bandage | High-risk, Silver Impregnated | High-risk, Negative-pressure Wound Vacuum | Total
Number analyzed (Participants) | 446 | 440 | 95 | 83 | 1064
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 446 | 440 | 95 | 83 | 1064
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 446 | 440 | 95 | 83 | 1064
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 66 | 14 | 12 | 159
  Not Hispanic or Latino | 379 | 374 | 81 | 71 | 905
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 85 | 79 | 17 | 14 | 195
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 183 | 185 | 40 | 36 | 444
  White | 178 | 176 | 38 | 33 | 425
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 446 | 440 | 95 | 83 | 1064
Enrollment Parameters [Count of Participants; unit: Participants] | 446 | 440 | 95 | 83 | 1064

OUTCOME MEASURES:

1. Primary Outcome: Infection Rate
Description: rate of post operative infection
Time Frame: 30 days from surgery
Measure: Count of Participants; unit: Participants
Groups:
- Low Risk, Border Bandage: low risk, (traditional) border bandage
Arm/Group | Low Risk, Silver Impregnated | Low Risk, Border Bandage | High-risk, Silver Impregnated | High-risk, Wound Vacuum
Number analyzed (Participants) | 446 | 440 | 95 | 83
Participants | 17 | 18 | 5 | 5

ADVERSE EVENTS:
Time Frame: 180-days post delivery (6-months)
Arm/Group | Low Risk, Silver Impregnated | Low Risk, Border Bandage | High-risk, Silver Impregnated | High-risk, Wound Vacuum
All-Cause Mortality (participants affected / at risk) | 0/446 | 0/440 | 0/95 | 0/83
Serious Adverse Events (participants affected / at risk) | 24/446 | 13/440 | 5/95 | 1/83
Other Adverse Events (participants affected / at risk) | 6/446 | 3/440 | 2/95 | 3/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Risk, Silver Impregnated (N=446) | Low Risk, Border Bandage (N=440) | High-risk, Silver Impregnated (N=95) | High-risk, Wound Vacuum (N=83)
POST-PARTUM HOSPITALIZATION (6-months) (Reproductive system and breast disorders) | 24 (29) | 13 (14) | 5 (7) | 1 (1) — INPATIENT HOSPITALIZATIONS (Post-partum) within 6-months of delivery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Risk, Silver Impregnated (N=446) | Low Risk, Border Bandage (N=440) | High-risk, Silver Impregnated (N=95) | High-risk, Wound Vacuum (N=83)
Superficial Wound Infections (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT04582045/Prot_SAP_000.pdf